CLINICAL TRIAL: NCT03228966
Title: Evaluating Indicators of Cardiac Function in Children Living With HIV in Western Kenya
Brief Title: Ped HIV - Echo Study: Kenya
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Duke Center for AIDS Research (Unknown); International AIDS Society (Other); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00083416
Record Dates: First submitted 2017-07-21; First posted 2017-07-25 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: HIV/AIDS; Cardiomyopathies
Keywords: Pediatric
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Cardiomyopathies | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma for viral load and inflammatory marker testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: Echocardiogram — Screening echocardiogram

SUMMARY:
Background: In children and adults living with HIV, cardiomyopathy is a major source of comorbidity. Traditional echocardiographic measures are insensitive and consequently cardiomyopathy often goes undiagnosed until late stages of disease. Myocardial deformation imaging represents a promising means to identify early dysfunction, but to date there have been no large studies using strain or strain rate to assess cardiac function in children with HIV and to establish predictors of worse cardiac function such as viral burden and ART regimen. These studies are critically important as earlier diagnosis and intervention represent the best means to alter the course of HIV-associated cardiomyopathy.

Objectives: To determine the association of biomarker levels, myocardial deformation, and viral load level history in HIV infected children attending Moi Teaching and Referral Hospital (MTRH) clinic.

Design: A cross-sectional study on clients attending HIV clinic, MTRH. Setting: Module 4 HIV clinic at MTRH in western Kenya, Africa. Population: HIV-infected children attending clinic in 2017 - 2018 Main Measures: Echocardiographic function assessment, Age, Immune status, other illnesses, ART status.

Conclusions: The study will explore the NIH/HIV High Priority Target area of HIV-associated cardiac co-morbidities and will enhance understanding of the relationship between cardiac function and viremia. The investigators expect to be able to reliably define a subset of children with worse cardiac function by risk factors: specific ART regimens, less time virally suppressed, and increased BNP biomarker.

DETAILED DESCRIPTION:
Research Summary:

1. Protocol Title: Evaluating Indicators of Cardiac Function in Children Living with Human Immunodeficiency Virus in Western Kenya
2. Purpose of Study: To determine the association of biomarker levels and relevant HIV history with cardiac function in HIV infected children attending Moi Teaching and Referral Hospital (MTRH) clinic.
3. Background & Significance:

   HIV-associated cardiomyopathy is a disease that exposes children with the infection to tremendous morbidity and mortality. Detection of cardiomyopathy is limited by traditional echocardiographic measures (i.e. left ventricular ejection fraction, LVEF), which do not detect cardiomyopathy until late stages of disease. Therefore, a critical need exists to determine HIV-associated cardiomyopathy risk through early detection. Prior to changes in traditional echocardiographic measures, newer cardiac imaging techniques such as myocardial deformation imaging (ie strain measurements) can detect decreased myocardial performance when LVEF is still normal. The lack of methods to detect early myocardial dysfunction and biomarkers that determine risk are major barrier for outcomes and treatment research.

   Myocardial deformation imaging represents a promising means to identify early dysfunction, but to date there have been no large studies using strain to assess cardiac function in children with HIV. Further, none have established predictors of worse cardiac function such as viral burden, immune status, zidovudine-containing ART regimens, and inflammatory state. This large-scale investigation utilizing the latest imaging techniques in evaluating cardiac function will provide first-in-kind data enabling estimation of prevalence of early HIV-associated cardiomyopathy as well as risk stratification. The study will explore the NIH/HIV High Priority Target area of HIV-associated cardiac co-morbidities and will enhance understanding of the relationship between cardiac function and viremia. Although these data will substantively enhance our understanding of early disease progression in children with subclinical HIV-associated cardiomyopathy, my long-term objective is to use these data in support of future work focused on early initiation of potentially, life altering therapies (such as angiotensin-converting enzyme inhibitor and digoxin medications) to children at highest risk for HIV-associated cardiac dysfunction in Africa and other resource poor regions of the world.

   The proposal objective is to determine the association of biomarker levels, myocardial deformation, and viral load level history in children with perinatally acquired HIV. Our central hypothesis is that risk of abnormal myocardial strain can be defined in terms of HIV clinical parameters - including viral load, antiretroviral therapy (ART), CD4 count, and serum biomarkers (such as b-natriuretic peptide, BNP). The investigators will accomplish our objectives with the following Specific Aims:

   AIM 1: Describe the prevalence of cardiomyopathy using myocardial deformation imaging compared with traditional echocardiographic measures in a large cohort of children living with HIV.

   Hypothesis 1: Strain and rate measurements will demonstrate presence of early cardiomyopathy not detected by traditional echocardiographic measures.

   AIM 2: Evaluate the association between HIV viral load and global longitudinal strain and strain rate.

   Hypothesis 2: Children with detectable replicating virus will have worse global longitudinal strain and strain rate measurements than those who are virally suppressed, and increasing viral load will be associated with worsening longitudinal strain and strain rate.

   AIM 3: Evaluate the association between b-natriuretic peptide level and myocardial strain.

   Hypothesis 3: There will be an inverse relationship between b-natriuretic peptide level and myocardial strain. The correlation between b-natriuretic peptide level and myocardial strain will potentially lead to screening thresholds in children living with HIV.
4. Design & Procedures:

The study will be a cross sectional design and conducted on consecutive HIV infected children seen in the AMPATH Pediatric HIV clinic whose mothers or caregivers give consent.

Each subject will undergo a 2-dimensional transthoracic echocardiogram after enrollment during her/his regularly scheduled clinic follow up as defined in the inclusion criteria. The echocardiogram will be completed with a portable cardiovascular ultrasound machine (GE Vivid q or similar) equipped with 4-8 MHz tissue-harmonic imaging probes. Images will be acquired with raw data and DICOM data at frame rates 60-100 frames/min. Additionally, electrocardiographic leads will be attached during image acquisition. The echocardiogram is anticipated to take less than 20 minutes of procedure time for the patient.

Traditional echocardiographic measurements will include LVEF, fractional shortening, and estimations of diastolic function such as mitral inflow E/A ratio. Additionally, assessment of the right ventricle will include indicators of pulmonary hypertension such as tricuspid regurgitant jet velocity, tricuspid valve annular plane systolic excursion (TAPSE), and pulmonary insufficiency end-diastolic gradient. Measurements will be performed according to American Society of Echocardiography standards. The definition of cardiomyopathy will be restricted to reduced left ventricular systolic function. Reduced left ventricular systolic function will be defined as ejection fraction less than 50% by traditional measures. Fractional shortening and myocardial deformation imaging (longitudinal strain) will be defined as reduced left ventricular systolic function if the value is less than 2 standard deviations below the published means for age.

Left ventricular global longitudinal strain and strain rate measurements will be made using the "length of line" technique from the apical 4-chamber, 2-chamber, and 3-chamber views. Right ventricular longitudinal strain and strain rate measurements will be made from the apical 4-chamber view using the same technique. All strain and strain rate measurements will be performed utilizing GE console analysis package (Netherlands) and TomTec ImageComTM software (Germany).

Data will be extracted from the electronic and paper medical record for key demographic and historical data including but not limited to markers of HIV infection (e.g., white blood cell counts, nadir and most recent CD4 counts, and HIV viral loads), duration since initiation of ART, type of regimen, regimen changes, lifetime ART exposure, anthropomorphic data (age, weight, height, sex, and gender), blood pressure measurements, and comorbidities.

Blood samples will be obtained as additional vials with the same clinically indicated venipuncture for all subjects. The primary study population will be children undergoing a routine clinically-indicated laboratory blood draw. However, children attending clinic for a routine follow up visit but not due for a laboratory blood draw will still be offered the opportunity to participate in the study as well. No more than 5 ml of blood will be drawn for the study. Children less than 3.5 kg will be excluded. The blood samples transported daily to the AMPATH Reference Laboratory at MTRH, which is accredited by the NIAID Division of AIDS. Samples will be labeled with study identification number only. The reference laboratory will be governed under the Duke - Moi Teaching and Referral Hospital data agreement. The investigators will analyze b-natriuretic peptide (BNP) levels for all subjects. Additionally, the remaining serum will be stored at the AMPATH Reference Laboratory for testing of inflammatory markers at Duke University. In order to understand mechanisms of cardiomyopathy in the HIV-infected, the investigators plan to secure additional funding to test markers of inflammation thought to be causative in cardiac dysfunction including: tumor necrosis factor alpha (TNF- α), interleukin (IL)-1b, IL-6, and IL-8. TNF- α, IL-1b, IL-6, and IL-8, and ST2. The investigators will store the blood specimens for up to 2 years after the last patient has been enrolled. Specimens will be destroyed or further IREC approval will be requested to maintain the stores beyond May 2020.

ELIGIBILITY:
Inclusion Criteria:

* Attending HIV care clinic for regular follow up visit
* < 14 years old
* Diagnosed HIV prior to age 10
* caregiver gives consent

Exclusion Criteria:

* unable to cooperate with echocardiogram

Ages: 1 Month to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children living with HIV attending regular scheduled follow up visit.
Sampling Method: Non-Probability Sample
Enrollment: 643 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Cardiac function inversely associated with HIV viral load | Day of clinic visit laboratory results
Cardiac function inversely associated with inflammatory marker levels | Day of clinic visit laboratory results
Cardiac function inversely associated with bio-marker levels | Day of clinic visit

CONTACTS AND LOCATIONS:
Overall Officials: Andrew W McCrary, MD, Principal Investigator — Duke University
Locations (1):
- Moi Teaching and Referral Hospital, Eldoret, Kenya

IPD SHARING:
Plan to Share IPD: Undecided